CLINICAL TRIAL: NCT02538341
Title: Safety and Effectiveness of Live Zoster Vaccine in Anti-TNF Users (VERVE Trial)
Brief Title: Safety and Effectiveness of Live Zoster Vaccine in Anti-Tumor Necrosis Factor (TNF) Users (VERVE Trial)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jeff Curtis, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VERVE-UM1; NCT01967316 (obsolete NCT alias); NCT02538757 (obsolete NCT alias)
Record Dates: First submitted 2015-08-18; First posted 2015-09-02 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis; Inflammatory Arthritis; Arthritis; Psoriatic Arthritis; Psoriasis; Ankylosing Spondylitis; Enteropathic Arthritis; Crohn's Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Arthritis, Psoriatic; Psoriasis; Spondylitis, Ankylosing; Crohn Disease | interventions — Vaccines; Herpes Zoster Vaccine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zostavax (Zoster Vaccine Live) (Active Comparator): Zostavax (zoster vaccine live) is used to prevent herpes zoster (HZ) virus (shingles) in people age 50 and older. Patients randomized to this arm will receive active herpes zoster (HZ) vaccine. It is administered as a single 0.65 mL dose subcutaneously in the deltoid region of the upper arm.
  Interventions: Biological: Herpes Zoster (HZ) Vaccine
- Placebo Normal Saline (Placebo Comparator): Saline injection: patients randomized to this arm will receive a single 0.65 mL dose subcutaneously in the deltoid region of the upper arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Herpes Zoster (HZ) Vaccine
  Other Names: Zostavax
  Arms: Zostavax (Zoster Vaccine Live)
Drug: Placebo
  Other Names: Normal Saline
  Arms: Placebo Normal Saline

SUMMARY:
The VaricElla zosteR VaccinE (VERVE) trial evaluates the safety and effectiveness of the Herpes zoster (HZ) vaccine for shingles, Zostavax, in patients over 50 years old with arthritis and other diseases who are using anti-tumor necrosis factor (TNF) therapy and who have not previously received the vaccine.

DETAILED DESCRIPTION:
Herpes zoster (HZ), also known as "shingles", is caused by reactivation and multiplication of the ubiquitous varicella zoster virus (VZV) that remains latent in everyone's sensory neurons following varicella, or "chickenpox". Among individuals who live to age 85, the lifetime risk for herpes zoster (HZ) is 50%, and more than one in five individuals affected by zoster develop post-herpetic neuralgia, resulting in chronic pain. Other serious complications include encephalitis, permanent vision loss, or more rarely, dissemination and death. Fortunately, a live attenuated vaccine is available and can reduce herpes zoster (HZ) risk by up to 70%. For patients with rheumatoid arthritis (RA), this vaccine has great potential to provide improved quality of life by reducing the incidence and complications associated with zoster. Due to the underlying disease and/or treatments (e.g. steroids) for rheumatoid arthritis (RA), the risk of herpes zoster (HZ) in rheumatoid arthritis patients is approximately double in the general population. This increased risk should make prevention of zoster and vaccination exceedingly important for rheumatoid arthritis patients. In fact, because of a higher overall absolute risk for herpes zoster (HZ) in rheumatoid arthritis, the vaccine yields a comparable or even greater absolute risk reduction to reduce the risk of shingles and post-herpetic neuralgia in a rheumatoid arthritis population as it does in the general population. However, the use of the herpes zoster (HZ) in rheumatoid arthritis, patients is very low (< 5%), and less frequently used than for the general population.

National guidelines from the Centers for Disease Control's (CDC) Advisory Committee on Immunization Practices (ACIP) recommend a single dose of the herpes zoster (HZ) vaccine for all individuals age 60 or older, with the vaccine more recently gaining Federal Drug Administration (FDA) -approval for administration to persons age 50 and older. While a large number of rheumatoid arthritis patients would otherwise be recommended to receive this vaccine on the basis of age, theoretical safety concerns related to vaccination likely explain the very low vaccination rates observed. Currently, the Federal Drug Administration (FDA), the Advisory Committee on Immunization Practices (ACIP), and the American College of Rheumatology (ACR) consider the live zoster vaccine contraindicated in patients receiving immunosuppressive medications, such as biologic therapies. Such contraindication stems from the theoretical safety concern that these individuals could develop a varicella-like infection from the vaccine virus strain. However, investigators hypothesize that this vaccine can safely be given in this setting, as no published data is available to suggest that these safety concerns are warranted. A growing body of observational data suggests that vaccinating rheumatoid arthritis patients receiving biologic therapies with this vaccine may in fact be safe. Moreover, and similarly with little or no evidence, the Advisory Committee on Immunization Practices (ACIP) considers the vaccine safe and acceptable for patients using methotrexate at doses commonly used to treat rheumatoid arthritis (e.g. <= 25mg/week) and for patients using glucocorticoids at prednisone-equivalent doses of ≤ 20 mg/day.

In light of 1) a substantial elevated herpes zoster (HZ) risk among rheumatoid arthritis patients; 2) national data showing most rheumatoid arthritis patients are not vaccinated for herpes zoster (HZ) ; and 3) the high effectiveness of this vaccine in the general population, the investigators propose to conduct the Varicella zostER VaccinE (VERVE) trial, a randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, and long-term effectiveness of the live herpes zoster (HZ) vaccine. This study will recruit 1,000 individuals age 50 years or older currently receiving anti-tumor necrosis factor (TNF) therapy for rheumatoid arthritis or other diseases. Within a relevant 6-week safety window, the investigators will collect serious adverse events (satisfying a regulatory definition of a Serious Adverse Event) including non-serious events of vaccine-strain varicella-like infection or herpes zoster (HZ). Beyond the key public health importance of the clinical question addressed, clinical trial methodological innovations anticipated for this unique large pragmatic trial. Additionally, the investigators will study vaccine tolerability and long-term effectiveness through a linkage to health plan data to allow for cost-effective follow-up while minimizing participant and study-site burden. Results from this study will facilitate the parent trial and change rheumatoid arthritis management by demonstrating the clinical safety and immunogenicity of the live zoster vaccine among current anti-tumor necrosis factor (TNF) users. Rheumatologists and other providers will be able to improve the care, outcomes, and quality of life for patients using anti-tumor necrosis factor (TNF) therapy, substantially decreasing the morbidity of herpes zoster and its complications over a lifetime.

ELIGIBILITY:
Inclusion Criteria:

* Must be 50 years of age or older
* Must be currently treated with an anti-tumor necrosis factor (TNF) therapy** at the time of study drug administration, allowing for small deviations in dosing frequency and logistic feasibility (e.g. study visits to occur on a week day). Date of previous dose of medication is required. Specifically, meets one of the following: Etanercept dose within 9 days (1 week + 2 days), Adalimumab dose within 16 days (2 weeks + 2 days), Certolizumab Subcutaneous (SC) dose within 16 to 32 days depending on frequency schedule (2 weeks + 2 days, or 4 weeks and 4 days), Golimumab Subcutaneous (SC) dose within 32 days (4 weeks + 4 days), Golimumab Intravenous (IV) dose within 64 days (9 weeks + 1 day), Infliximab IV dose within last 64 days (9 weeks + 1 day)

  **any form of biosimilar for the above listed anti-tumor necrosis factor (TNF) medications is acceptable
* Diagnosis of rheumatoid arthritis or another inflammatory arthritis (Phase 1A); or other inflammatory condition (e.g. psoriasis) requiring use of anti-tumor necrosis factor (TNF) therapy (Phase 1B and II)
* Phase I subjects must test positive for varicella-zoster virus (VZV) antibody immunoglobulin G (IgG)
* Subjects should have a self-reported history of prior varicella infection (i.e. chicken pox) or long-term residence (>30 years) in the continental United States.
* Phase IA subjects must not have received any oral or systemic glucocorticoids within 30 days prior to vaccination. Intra-articular glucocorticoid injections and inhaled glucocorticoids within the previous 30 days are acceptable.
* Subjects should be on stable doses of all biologic and non-biologic Disease-modifying antirheumatic drugs (DMARDs) for a minimum of 30 days prior to vaccination.
* Eligible women must be post-menopausal (> 1 year since last menstrual period) or have a surgical history of bilateral oophorectomy or hysterectomy.
* Subjects should be ambulatory, community dwelling and capable of giving informed consent.

Exclusion Criteria:

* Documented varicella-zoster virus (VZV) antibody immunoglobulin G (IgG) negative result
* Prior use of the zoster vaccine (Zostavax®, Merck)
* Glucocorticoids at a prednisone-equivalent daily dose > 10mg/day (for Phase 1B and Phase II participants; all systemic glucocorticoid use is prohibited for Phase 1A patients)
* Any known contraindication to Zostavax® vaccine, including allergy or sensitivity to gelatin or any other vaccine component
* Known human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS)
* Currently receiving radiation or chemotherapy for any type of malignancy
* Any current use (within the last 30 days) of acyclovir, valacyclovir, famciclovir, or foscarnet
* Receipt of any other immunizations within one month before study vaccination (2 weeks in the case of inactivated influenza vaccines or other non-replicating immunization products [e.g., diphtheria-tetanus (dT), pneumococcal vaccine, hepatitis A vaccine, hepatitis B vaccine]), or scheduled within 6 weeks after recruitment.
* Active infection or inter-current illness (e.g., urinary tract infection, influenza)
* Participated in an investigational study within 1 month prior to study entry
* Active drug or alcohol use, dependence, or any other reason that, in the opinion of the site investigator, would interfere with the study
* Significant underlying illness that would be expected to prevent completion of the study (e.g., life-threatening disease likely to limit survival to less than 3 years)
* Any other reason that, in the opinion of the site investigator, would interfere with required study related evaluations (e.g. uncontrolled comorbidity, life expectancy < 1 year)
* Patients who have household contact with varicella-susceptible pregnant women or severely immunosuppressed individuals without history of primary varicella.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Curtis, MD, MS, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (34):
- United States (34):
  - Rheumatology Associates, PC, Birmingham, Alabama
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Clinical and Translational Research Center of Alabama, PC, Tuscaloosa, Alabama
  - SunValley Arthritis Center, Ltd, Peoria, Arizona
  - Arthritis Association of Southern California, Los Angeles, California
  - The Regents of the University of California Los Angeles, Los Angeles, California
  - Rheumatology Consultants of Delaware dba Delaware Arthritis, Lewes, Delaware
  - Center for Arthritis and Rheumatic Diseases, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Arthritis Research of Florida, Inc, Palm Harbor, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - West Broward Rheumatology Associates, Inc, Tamarac, Florida
  - North Georgia Rheumatology Group, Lawrenceville, Georgia
  - Arthritis Research Center Foundation, NDB, Wichita, Kansas
  - Ochsner Clinic Baton Rouge, Baton Rouge, Louisiana
  - Ochsner Clinic Foundation, New Orleans, New Orleans, Louisiana
  - Rheumatology & Osteoporosis Specialists, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Pine Hollow Partners, East Lansing, Michigan
  - St. Paul Rheumatology, Eagan, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - The Center for Rheumatology, LLP, Albany, New York
  - Mary Imogene Bassett Hospital, Bassett Research Institute, Cooperstown, New York
  - The Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Carolina Health Specialists, Myrtle Beach, South Carolina
  - Arthritis Associates, PLLC, Hixson, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - West Virginia Research Institute, PLLC, South Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Curtis JR, Cofield SS, Bridges SL Jr, Bassler J, Deodhar A, Ford TL, Huffstutter J, Jankeel A, Kivitz A, Kamal S, Lindsey S, Messaoudi I, Mendoza N, Michaud K, Mikuls TR, Ridley D, Shergy W, Siegel SAR, Winthrop KL. The Safety and Immunologic Effectiveness of the Live Varicella-Zoster Vaccine in Patients Receiving Tumor Necrosis Factor Inhibitor Therapy : A Randomized Controlled Trial. Ann Intern Med. 2021 Nov;174(11):1510-1518. doi: 10.7326/M20-6928. Epub 2021 Sep 28. PMID 34570596

RESULTS

PARTICIPANT FLOW:
Groups:
- Zoster Vaccine Live (Zostavax): Zostavax (zoster vaccine live) is used to prevent herpes zoster virus (shingles) in people age 50 and older. Patients randomized to this arm will receive active Herpes Zoster Vaccine. It is administered as a single 0.65 mL dose subcutaneously in the deltoid region of the upper arm.
  Herpes Zoster Vaccine
- Placebo Normal Saline: Saline injection: patients randomized to this arm will receive a single 0.65 mL dose subcutaneously in the deltoid region of the upper arm.
  Placebo
Period: Overall Study
Arm/Group | Zoster Vaccine Live (Zostavax) | Placebo Normal Saline
Started | 310 | 307
Week 6 (Primary Outcome) | 303 | 299
Month 6 (Safety Outcome) (All participants were followed in a blinded manner until Month 6 when clinical sites and participants were unblinded. Participants randomized to placebo completed the study at Month 6.) | 276 | 260
1 Year Visit (As an exploratory outcome to assess the immunologic persistence of live herpes zoster vaccine among participants randomized to the vaccine, only those participants were invited to provide a Year 1 blood sample for the same lab assessments.) | 254 | 0
Completed | 254 | 260
Not Completed | 56 | 47
Not completed — Lost to Follow-up | 51 | 46
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoster Vaccine Live (Zostavax) | Placebo Normal Saline | Total
Number analyzed (Participants) | 310 | 307 | 617
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 62.7 (7.6) | 63.1 (7.4) | 62.9 (7.5)
Age, Customized [Count of Participants; unit: Participants]
  Age: 50-59 | 126 | 102 | 228
  Age: 60-69 | 125 | 142 | 267
  Age: 70-79 | 50 | 55 | 105
  Age: 80-89 | 9 | 7 | 16
  Age: 90-99 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 201 | 408
  Male | 103 | 106 | 209
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 14 | 38
  White | 202 | 197 | 399
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 81 | 91 | 172
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 14 | 12 | 26
  Ethnicity: Not Hispanic | 208 | 194 | 402
  Ethnicity: Other Ethnicity | 7 | 7 | 14
  Ethnicity: Unknown/ Not reported | 81 | 94 | 175
Region of Enrollment [Number; unit: participants]
  United States | 310 | 307 | 617

OUTCOME MEASURES:

1. Primary Outcome: GMFR (Geometric Mean Fold Rise ) in Varicella Zoster Virus (VZV) Glycoprotein Enzyme-linked Immunosorbent Assay (gpELISA) Immunoglobulin G (IgG) Levels From Baseline at 6 Weeks
Description: Study protocol defined measure for immunogenicity samples.
Time Frame: 6 weeks post vaccination
Population: Zoster vaccine live arm 7 did not complete Week 6; 5 lost to follow-up, 2 withdrew consent. Placebo arm 8 did not complete Week 6; 5 lost to follow-up, 3 withdrew consent. Zoster vaccine live arm 300 immunogenicity samples collected, 294 useable immunoglobulin G (IgG) samples, 287 usable immunoglobulin G (IgG) sample pairs. For the placebo arm 298 immunogenicity samples collected, 289 useable immunoglobulin G (IgG) samples, 259 usable immunoglobulin G (IgG) sample pairs.
Measure: Geometric Mean (95% Confidence Interval); unit: GMFR (Geometric Mean Fold Rise )
Units Other Than Participants: IgG samples pairs
Arm/Group | Zoster Vaccine Live (Zostavax) | Placebo Normal Saline
Number analyzed (Participants) | 303 | 299
Number analyzed (IgG samples pairs) | 287 | 289
GMFR (Geometric Mean Fold Rise ) | 1.33 [1.17 to 1.51] | 1.02 [0.91 to 1.14]
Statistical Analysis 1: Comparison: Zoster Vaccine Live (Zostavax) vs Placebo Normal Saline; Study protocol defined measure for immunogenicity samples. Participants must have at least 1 post vaccine immunogenicity measure to determine the GMFR (a priori analysis); Test type: Other; p = 0.0023, a generalized linear model — p values, from a generalized linear model on the rank order of the week 6 - baseline change using normal distribution and reciprocal link; p value,from a generalized linear model on the rank order of the week 6 - baseline change using normal distribution and reciprocal link

2. Primary Outcome: GMFR (Geometric Mean Fold Rise ) in Varicella Zoster Virus (VZV) Enzyme-linked Immune Absorbent Spot (ELISpot) Interferon Gamma (IFNg) Levels From Baseline at 6 Weeks
Description: Study protocol defined measure for immunogenicity samples.
Time Frame: 6 weeks post vaccination
Population: Zoster vaccine live arm 7 did not complete Week 6; 5 lost to follow-up, 2 withdrew consent. Placebo arm 8 did not complete Week 6; 5 lost to follow-up, 3 withdrew consent. For the zoster vaccine live arm 300 immunogenicity samples collected, 290 useable interferon gamma (IFNg) samples, 259 usable interferon gamma (IFNg) sample pairs. For the placebo arm 298 immunogenicity samples collected, 289 useable interferon gamma (IFNg) samples, 275 usable interferon gamma (IFNg)sample pairs.
Measure: Geometric Mean (95% Confidence Interval); unit: GMFR (Geometric Mean Fold Rise )
Units Other Than Participants: lab samples pairs
Arm/Group | Zoster Vaccine Live (Zostavax) | Placebo Normal Saline
Number analyzed (Participants) | 303 | 299
Number analyzed (lab samples pairs) | 259 | 275
GMFR (Geometric Mean Fold Rise ) | 1.39 [1.07 to 1.82] | 1.15 [0.88 to 1.50]
Statistical Analysis 1: Comparison: Zoster Vaccine Live (Zostavax) vs Placebo Normal Saline; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.31, a generalized linear model — [p-value comment as in outcome 1, analysis 1]; p values, from a generalized linear model on the rank order of the week 6 - baseline change using normal distribution and reciprocal link

3. Secondary Outcome: GMFR (Geometric Mean Fold Rise ) in Varicella Zoster Virus (VZV) Glycoprotein Enzyme-linked Immunosorbent Assay (gpELISA) Immunoglobulin G (IgG) Levels From Baseline at 1 Year
Description: Study defined measure from labs. GMFR (Geometric Mean Fold Rise ) in varicella zoster virus (VZV) glycoprotein enzyme-linked immunosorbent assay (gpELISA) immunoglobulin G (IgG) levels
Time Frame: Baseline to 1 year
Population: Zoster vaccine live arm 56 did not complete Year 1; 51 lost to follow-up, 3 withdrew consent, 2 deaths prior to month 6. Vaccine arm only. Placebo arm not applicable for this exploratory outcome. For the zoster vaccine live arm 131 immunogenicity samples collected, 122 useable immunoglobulin G (IgG) samples, 114 usable immunoglobulin G (IgG) sample pairs.
Measure: Count of Units; unit: lab samples
Units Other Than Participants: lab samples
Arm/Group | Zoster Vaccine Live (Zostavax)
Number analyzed (Participants) | 254
Number analyzed (lab samples) | 114
lab samples
  ≤ Baseline | 41
  Within 20% | 6
  > 20% | 67

4. Secondary Outcome: GMFR (Geometric Mean Fold Rise ) in Varicella Zoster Virus (VZV) Enzyme-linked Immune Absorbent Spot (ELISpot) Interferon Gamma (IFNg) Levels From Baseline at 1 Year
Description: Study defined measures from labs. GMFR (Geometric Mean Fold Rise ) in Varicella Zoster Virus (VZV) enzyme-linked immune absorbent spot (ELISpot) interferon gamma (IFNg)
Time Frame: Baseline to 1 year
Population: Zoster vaccine live arm 56 did not complete Year 1; 51 lost to follow-up, 3 withdrew consent, 2 deaths prior to month 6. Vaccine arm only. Placebo arm not applicable. For the zoster vaccine live arm 131 immunogenicity samples collected, 125 useable interferon gamma (IFNg) samples, 116 usable interferon gamma (IFNg) sample pairs.
Measure: Count of Units; unit: lab samples
Units Other Than Participants: lab samples
Arm/Group | Zoster Vaccine Live (Zostavax)
Number analyzed (Participants) | 254
Number analyzed (lab samples) | 116
lab samples
  ≤ Baseline | 87
  Within 20% | 2
  > 20% | 27

5. Secondary Outcome: Number of Samples With Confirmed Varicella
Description: Evaluated all serious adverse events (SAEs) AND non-serious varicella zoster virus (VZV) events
Time Frame: "Placebo Normal Saline Arm/Group was assessed up to 6 months and the "Zoster Vaccine Live (Zostavax)" Arm/Group was assessed up to 1 year
Population: Lab samples collected for testing for varicella
Measure: Number; unit: lab sample
Units Other Than Participants: lab sample
Arm/Group | Zoster Vaccine Live (Zostavax) | Placebo Normal Saline
Number analyzed (Participants) | 310 | 307
Number analyzed (lab sample) | 4 | 4
lab sample
  Total Samples Tested | 4 | 4
  Total Sample with Confirmed Varicella | 0 | 0

6. Secondary Outcome: Vaccine Tolerability Within 42 Days Following Vaccination.
Description: Patient self report data in the form of a diary to include injection site reactions; symptoms of swelling, redness or tenderness. Diary was completed from study injection administration up to 6 week visit
Time Frame: 42 days post vaccination
Population: 7 participants from the Zostavax arm and 8 participants from the placebo arm did not complete 6 week visit for various a reasons (e.g., lost to follow up, consent withdrawn , etc.)
Measure: Count of Participants; unit: Participants
Arm/Group | Zoster Vaccine Live (Zostavax) | Placebo Normal Saline
Number analyzed (Participants) | 303 | 299
Participants | 60 | 13

7. Secondary Outcome: Evaluate Rheumatoid Arthritis Disease Activity Using the Clinical Disease Activity Index (CDAI)
Description: Rheumatoid arthritis disease activity will be measured using the clinical disease activity index (CDAI). Clinical disease activity index (CDAI) is a measure of rheumatoid arthritis disease activity and is scored on a scale ranging from 0-76, with lower numbers indicated better control of disease. Values <=10 are consistent with low disease activity or remission.
Time Frame: 42 days post vaccination
Population: 120 participants on Zostavax arm and 129 participants on placebo arms were non-rheumatoid arthritis participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Zoster Vaccine Live (Zostavax) | Placebo Normal Saline
Number analyzed (Participants) | 190 | 178
score on a scale
  CDAI at Baseline | 9.54 (10.6) | 9.34 (9.77)
  CDAI at week 6 | 10.48 (10.93) | 10.31 (10.87)
  Changes in CDAI | 0.77 (7.33) | 0.98 (8.55)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events (SAEs) within 42 days of vaccination (placebo and vaccine). 6 months (final safety assessment for placebo arm).Serious Adverse Events (SAEs) up to 1 year (final safety assessment for treatment arm).
Description: Serious adverse events (SAEs) AND non-serious varicella zoster virus events. SAEs will include all that satisfy the FDA-accepted definition of SAEs (results in death, life threatening, results in or prolongs hospitalization, and any Herpes Zoster event). Adverse events (non-serious) include rashes,blisters,fever of greater than 101,sickness/illness. Also, any redness, swelling, tenderness of the injection site or any other body part.
Arm/Group | Zoster Vaccine Live (Zostavax) | Placebo Normal Saline
All-Cause Mortality (participants affected / at risk) | 3/310 | 0/307
Serious Adverse Events (participants affected / at risk) | 10/310 | 8/307
Other Adverse Events (participants affected / at risk) | 120/310 | 75/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoster Vaccine Live (Zostavax) (N=310) | Placebo Normal Saline (N=307)
Ductal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pseudoseizures (Nervous system disorders) | 1 (1) | 0 (0)
Syncope and collapse (Nervous system disorders) | 0 (0) | 1 (1)
Blocked Bowel (Gastrointestinal disorders) | 3 (3) | 0 (0)
Respiratory Syncytial Virus Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis due to pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Right groin pain secondary to edema of the right hip adductor (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 0 (0)
Left Ureteral Obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Elevated blood pressure (Vascular disorders) | 0 (0) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Death (Congenital, familial and genetic disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoster Vaccine Live (Zostavax) (N=310) | Placebo Normal Saline (N=307)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eye pain/Redness (Eye disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 14 (14) | 11 (14)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 47 (61) | 7 (13)
Infection (Infections and infestations) | 8 (15) | 9 (18)
Anaphylaxis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (General disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bug Bites (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fever, Flu like Symptom (General disorders) | 9 (10) | 8 (12)
Nausea (Gastrointestinal disorders) | 4 (6) | 1 (2)
Psoriasis Flare (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Ankle Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthritis pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Chelitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Cold (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (General disorders) | 1 (1) | 1 (1)
Edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot and Groin Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Headache , Migraine (General disorders) | 2 (2) | 3 (3)
Sore Throat (General disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poison Ivy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ruptured vericose vein (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sprained ankle (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Angiomyolipoma (Renal and urinary disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 1 (1) | 0 (0)
Cat Bite (General disorders) | 1 (1) | 0 (0)
Heart Irregularities (Cardiac disorders) | 0 (0) | 1 (1)
Herpes sore (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bursitis (Infections and infestations) | 0 (0) | 1 (1)
Canker sore (General disorders) | 0 (0) | 1 (1)
hidradenitis (General disorders) | 0 (0) | 1 (1)
Low Blood Sugar (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lower Extremity Pain (General disorders) | 0 (0) | 1 (1)
Law Pain (General disorders) | 0 (0) | 1 (1)
Not Specifies (General disorders) | 20 (24) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT02538341/Prot_SAP_000.pdf